CLINICAL TRIAL: NCT01755897
Title: A Multicenter, Prospective, Randomized Trial of Adjuvant Chemotherapy for Early-Stage Cervical Cancer Patients
Acronym: CC-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Zhejiang University (Other); Shandong University (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of Department of Gynecology and Obstetrics, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSEM GOG-002; 2012-GYN/CC-01 (Other: Tongji Hospital, HUST)
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer; Uterine Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant Chemotherapy (Arm A) (Experimental): Paclitaxel (T): 135-175 mg/m(2) intravenously (IV) on day 1, administrated intravenously over 3 hours; followed by cisplatin 75-85 mg/m(2) IV on day 2 and 3. Patients received at least 3 cycles at 4-week intervals beginning 2-3 weeks after surgery. 3-6 cycles as necessary.
  Interventions: Procedure: radical hysterectomy + pelvic lymph node dissection; Drug: Paclitaxel; Drug: Cisplatin
- Concurrent radiochemotherapy, CCRT (Arm B) (Active Comparator): Pelvic RT is delivered using IMRT technique, 45～50.4 Gy/4～7 weeks, brachytherapy will been given as necessary. Cisplatin 35 mg/m(2) IV once a week. Total treatment time is 6-7 weeks.
  Interventions: Procedure: radical hysterectomy + pelvic lymph node dissection; Drug: Cisplatin; Radiation: Pelvic RT

INTERVENTIONS:
Procedure: radical hysterectomy + pelvic lymph node dissection
Drug: Paclitaxel — 135-175 mg/m(2) intravenously (IV) on day 1
  Arms: Adjuvant Chemotherapy (Arm A)
Drug: Cisplatin — 75 mg/m(2) IV on day 2 and 3
  Arms: Adjuvant Chemotherapy (Arm A)
Drug: Cisplatin — 35 mg/m(2) IV once a week
  Arms: Concurrent radiochemotherapy, CCRT (Arm B)
Radiation: Pelvic RT — IMRT
  Arms: Concurrent radiochemotherapy, CCRT (Arm B)

SUMMARY:
We will conduct a trial to determine whether paclitaxel/cisplatin (TP) as an adjuvant chemotherapy after radical surgery improve disease-free survival (DFS) and overall survival (OS), as well as the quality of life (QoL) among early-stage (FIGO stage IB-IIA) cervical cancer patients with risk factors.

ELIGIBILITY:
Inclusion Criteria:

* FIGO stage: ⅠB～ⅡA, cervical cancer;
* Age≤60 years; female, Chinese women;
* Initial treatment is radical hysterectomy + pelvic lymph node dissection;
* Pathological diagnosis: cervical squamous cell invasive carcinoma;
* Pathologic examination and meet the following one of the indications of adjuvant therapy: ① lymph node metastasis, ② parametrial invasion, ③ ≥ 2/3 deep stromal invasion, ④ histopathological grading in poorly differentiated (G2 to G3), ⑤ lymphatic vascular space involvement, ⑥ tumor diameter> 4cm;
* Laboratory tests: WBC≥4×10(9)/L, NEU≥2×10(9)/L, PLT≥80×10(9)/L, serum bilirubin≤ 1.5 times the upper limit of normal, transaminase≤ 1.5 times the upper limit of normal, BUN, Cr≤ normal
* Performance status: Karnofsky score≥60;
* No prior treatment;
* Receiving extensive resection of uterus (type III) plus pelvic lymph nodes wide resection; pathologically diagnosed with cervical squamous cell carcinoma;
* Provide written informed consent.

Exclusion Criteria:

* With severe or uncontrolled internal disease, unable to receive surgery and/or unsuitable for radiotherapy or chemotherapy
* History of organ transplantation, immune diseases;
* History of serious mental illness, a history of brain dysfunction;
* Drug abuse or a history of drug abuse;
* Suffering from other malignancies;
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) | up to 3-year
  DFS was definite as the time from randomization to disease recurrence (including death from recurrence if it was the first manifestation of recurrence), death without recurrence.

SECONDARY OUTCOMES:
3-year overall survivals (OS) | 3-year
Quality of Life in two arms | 3 years
chemotherapy- and radiotherapy- related adverse effects respectively in two arms | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD, PhD, Study Chair — Huazhong University of Science and Technology
Locations (3):
- China (3):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Background] Weng D, Xiong H, Zhu C, Wan X, Chen Y, Wang X, Zhang Y, Jiang J, Zhang X, Gao Q, Chen G, Xing H, Wang C, Li K, Chen Y, Mao Y, Hu D, Pan Z, Chen Q, Cui B, Song K, Yi C, Peng G, Han X, An R, Fan L, Wang W, Xiong T, Chen Y, Tang Z, Li L, Yang X, Cheng X, Lu W, Wang H, Kong B, Xie X, Ma D. Adjuvant chemotherapy versus adjuvant concurrent chemoradiotherapy after radical surgery for early-stage cervical cancer: a randomized, non-inferiority, multicenter trial. Front Med. 2023 Feb;17(1):93-104. doi: 10.1007/s11684-021-0892-z. Epub 2022 Nov 23. PMID 36422763